CLINICAL TRIAL: NCT01133964
Title: Dairy Proteins and Postprandial Appetite Regulation and Energy Expenditure
Acronym: MAES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Janne Kunchel Lorenzen, Cand. Scient., Department of Human Nutrition, Life, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B256
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2008-09

CONDITIONS: Obesity
Keywords: Dairy proteins; Appetite regulation; Energy expenditure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- milk (Experimental): skim milk
  Interventions: Dietary Supplement: dairy proteins
- casein drink (Experimental)
  Interventions: Dietary Supplement: dairy proteins
- whey drink (Experimental)
  Interventions: Dietary Supplement: dairy proteins
- water (Sham Comparator)
  Interventions: Dietary Supplement: dairy proteins

INTERVENTIONS:
Dietary Supplement: dairy proteins — Protein drinks with 3.5% protein. The protein source will be whey, casein or whey and casein (20:80; normal content in the milk). In the arm with water no protein will be added.

SUMMARY:
The aim of this study is to examine the effect of dairy proteins (whey and casein) on postprandial appetite regulation and energy expenditure.

DETAILED DESCRIPTION:
Several studies have shown that a high protein intake is associated with a increased loss of body weight and body fat as compared to a diet with a normal or low protein content. The effect seems to be due to a higher diet induced thermogenesis and increase satiety.

Milk has a high content of proteins. It contains two very different types of protein: whey and casein. Whey is a soluble protein whereas casein clots into the stomach, which delays its gastric emptying and thus probably results in a slower release of amino acids. It is therefore very likely that the two types of protein affect the thermogenesis and appetite regulation differently.

The aim of the present study is to examine the effect of dairy proteins (whey and casein) on postprandial energy expenditure, substrate oxidation and appetite regulation.

The study will have a cross-over design including four meals each including a test drink (milk, casein drink, whey drink or water).

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* body mass index (BMI) 25-30 kg/m2
* 18-50 years
* weight stable

Exclusion Criteria:

* smoker
* regular use of medicine
* elitist athletes
* participation in other intervention studies

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Subjective appetite sensation | 5 hours
Energy expenditure | 5 hours
Substrate oxidation | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Dr., Principal Investigator — Department of Human Nutrition, Life, University of Copenhagen
Locations (1):
- Department og Human Nutrition, Life, University of Copenhagen, Copenhagen, Denmark